CLINICAL TRIAL: NCT01407302
Title: Optimal Head Rotation and External Landmark for Internal Jugular Vein Cannulation After Placement of Proseal Laryngeal Mask Airway
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Gwak Mi Sook, Professor, Samsung Medical Center
Other Study IDs: 2011-04-024
Record Dates: First submitted 2011-07-21; First posted 2011-08-02 (Estimated); Last update posted 2013-12-25 (Estimated); Status verified 2013-12

CONDITIONS: General Anesthesia With Laryngeal Mask Airway (LMA)
Keywords: Laryngeal mask airway; internal jugular vein cannulation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- LMA group: patients undergoing general anesthesia with LMA insertion
  Interventions: Other: Head rotation
- E-tube group: patients undergoing general anesthesia with e-tube
  Interventions: Other: Head rotation

INTERVENTIONS:
Other: Head rotation — Repeated ultrasonographic examination according to the degree of head rotation (examination of overlap index of internal jugular vein and common carotid artery, and accuracy of external landmark of jugular cannulation)

SUMMARY:
Recently, laryngeal mask airway (LMA) placements are frequently performed for general anesthesia. The investigators occasionally encounter a clinical situation to perform internal jugular vein (IJV) cannulation after LMA insertion, especially for difficult airway in subjects undergoing major surgery. However, anatomic relations of IJV and common carotid artery (CCA) in patient with LMA placement have been reported to be different from those in patients with endotracheal tube. The degree of overlapping of the right IJV and CCA after LMA placement was greater than before LMA placement. Furthermore, there are many cases of complete overlapping right IJV and CCA after LMA placement. Therefore, the risk of puncturing CCA increases when the investigators try to cannulate IJV after LMA placement. Furthermore, the central landmark commonly used for IJV cannulation was proved to show low success rate after LMA placement in previous report.

The investigators carefully examined the anatomic relations of IJV and CCA after LMA insertion with ultrasonography, and found that the degree of overlapping is different according to the degree of head rotation. The investigators postulated that if the degree of overlapping is different according to the degree of head rotation after LMA insertion, the investigators can find the angle of head rotation for least overlapping and reduce the risk of CCA puncture. Therefore, the investigators tried (1) to find the optimal head rotation angle appropriate for puncturing IJV after LMA placement, and (2) to find suitable landmark adequate for IJV cannulation after LMA placement.

DETAILED DESCRIPTION:
Recently, laryngeal mask airway (LMA) placements are frequently performed for general anesthesia. The investigators occasionally encounter a clinical situation to perform internal jugular vein (IJV) cannulation after LMA insertion, especially for difficult airway in subjects undergoing major surgery. However, anatomic relations of IJV and common carotid artery (CCA) in patient with LMA placement have been reported to be different from those in patients with endotracheal tube. The degree of overlapping of the right IJV and CCA after LMA placement was greater than before LMA placement. Furthermore, there are many cases of complete overlapping right IJV and CCA after LMA placement. Therefore, the risk of puncturing CCA increases when the investigators try to cannulate IJV after LMA placement. Furthermore, the central landmark commonly used for IJV cannulation was proved to show low success rate after LMA placement in previous report. Previous study recommended the lower puncture point near that area where the clavicular head of the sternocleidomastoid muscle attaches to the clavicle, because CCA was not observed in the vicinity of the IJV after LMA insertion. Even though they performed test puncture at the lower puncture point in 20 patients and found no complications, the lower puncture point is not the usual site for IJV cannulation for most anesthesiologists. It is known that increased head rotation is associated with high probability of CCA contact. The investigators carefully examined the anatomic relations of IJV and CCA after LMA insertion with ultrasonography, and found that the degree of overlapping is different according to the degree of head rotation. The investigators postulated that if the degree of overlapping is different according to the degree of head rotation after LMA insertion, the investigators can find the angle of head rotation for least overlapping and reduce the risk of CCA puncture. Therefore, the investigators tried (1) to find the optimal head rotation angle appropriate for puncturing IJV after LMA placement, and (2) to find suitable landmark adequate for IJV cannulation after LMA placement.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing general anesthesia with laryngeal mask airway insertion

Exclusion Criteria:

* patients undergoing emergency surgery
* patients with anatomical problem of airway
* anticipated difficult airway
* patients with hemodynamic unstability
* patients with severe cardiopulmonary disease

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing general anesthesia with laryngeal mask airway insertion
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2011-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
overlap index | at 5 min after anesthesia induction
  The overlap index was derived from the ratio of the overlapping length of the IJV to the horizontal diameter of the CCA measured on the ultrasonographic image. The formula of calculation is as follows: overlap index = [overlap length (mm)/ CCA diameter (mm)] X 100(%), the measurements were repeated according to the degree of head rotation (neutral, 15 degree, 30 degree, 45 degree)

SECONDARY OUTCOMES:
The success of simulated internal jugular vein puncture (central landmark) | at 5 min after anesthesia induction
  The success of internal jugular vein puncture guided by the central landmark simulated on the ultrasonographic images, the measurements were repeated according to the degree of head rotation (neutral, 15 degree, 30 degree, 45 degree)
The success of simulated internal jugular vein puncture (external jugular vein landmark) | at 5 min after anesthesia induction
  The success of internal jugular vein puncture as guided by 1.5 cm or 2.5 cm medial to the external jugular vein simulated on the ultrasonographic images, the measurements were repeated according to the degree of head rotation (neutral, 15 degrees, 30 degrees, 45 degrees)

CONTACTS AND LOCATIONS:
Overall Officials: Mi Sook Gwak, M.D.,Ph.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea